CLINICAL TRIAL: NCT00325975
Title: Immune Responses to Vaccinia Virus Vaccination
Brief Title: Immune Responses to Smallpox Vaccination
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030090; 03-I-0090
Record Dates: First submitted 2006-05-15; First posted 2006-05-15 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-03-15

CONDITIONS: Smallpox Vaccine
Keywords: Smallpox; Variola; Orthopoxvirus; Virus; Immunogenicity; Smallpox Vaccine
MeSH Terms: conditions — Smallpox; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
This study will examine how people s immune systems respond to inoculation with vaccinia virus the standard vaccine used to protect against smallpox and how these responses correlate with symptoms they develop after receiving the vaccine.

People 18 years of age and older who are scheduled to receive smallpox vaccination as a routine part of their employment (e.g., laboratory worker, health care worker, or emergency response worker) may be eligible for this study. They may or may not have been vaccinated previously. In addition, individuals who were vaccinated against smallpox at least 6 months before starting the study may participate as control subjects. All candidates will be screened with a brief medical history and physical examination.

Participants in the following vaccination categories will undergo the procedures described for their group:

Vaccine Recipient Frequent Follow-up

Participants will come to the NIH Clinical Center every 2 to 3 days for a total of 7 visits over a 2-week period. At each visit, starting the day of vaccination, they will have the following procedures:

* Brief skin examination, possibly with photographs of skin lesions;
* Throat and skin swabs for vaccinia virus culture;
* Blood draw (about 8 teaspoonfuls).

Additional blood samples will be collected 1 month after vaccination and again within a year after vaccination. The blood will be analyzed for the immune response to the vaccine, genetic differences that might influence differences in immune response, and the presence of vaccinia virus.

Participants will fill out a diary card every day for 3 weeks after vaccination to record any symptoms. Individuals who develop symptoms lasting more than 2 weeks, such as persistent or new skin lesions, will return to the clinic for additional skin exams and blood tests. Individuals who develop vaccine side effects may have a urine culture for vaccinia virus.

Vaccine Recipient Infrequent Follow-up

Participants will come to the NIH Clinical Center for blood tests on the day of vaccination, 4 weeks after vaccination, and once again within a year after vaccination. At each visit, 6 teaspoonfuls of blood will be drawn. This group will also include individuals who have been vaccinated within 8 months of entering the study and are not currently receiving the vaccine, but for whom blood samples are not available.

Control Group Vaccinated at Least 6 Months Before Entering the Study

Participants will come to the NIH Clinical Center for blood tests every 2 to 3 days for 2 weeks, then at 1 month after the first blood draw, and again within a year of the first blood draw. About 8 teaspoonfuls of blood will be drawn at each visit.

DETAILED DESCRIPTION:
Vaccinia virus is used to vaccinate persons to prevent disease with smallpox. Limited information is available regarding cellular immune responses to vaccinia virus. We will obtain blood from vaccinated persons and measure immune responses in vitro to the virus and correlate these findings with symptoms from vaccination. Elucidation of these responses might help to predict side effects associated with vaccination, and suggest new therapies to reduce these side effects.

ELIGIBILITY:
* INCLUSION CRITERIA:

  18 years of age or older

Both males and females

Patients will be checked on day 0 and those with a hemoglobin of greater than or equal to12 g/dL will have blood drawn as described in the protocol. Patients with a hemoglobin of 11-11.9 will have a 50% reduction in the amount of blood drawn after the first visit from 40 ml per visit to 20 ml per visit. Patients with a hemoglobin less than 11 g/dL will be terminated from the study and referred for medical follow-up.

Able to sign the consent form and be willing to comply with study procedures.

Must be a laboratory worker, health care worker, or emergency response worker who is receiving smallpox vaccination as a routine part of employment. Persons who were previously vaccinated at least 8 months ago are eligible.

EXCLUSION CRITERIA:

Active substance abuse or history of prior substance abuse that may interfere with protocol compliance or compromise patient safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2003-02-04; Study Completion 2016-03-15

PRIMARY OUTCOMES:
Vaccinia virus is used to vaccinate persons to prevent disease with smallpox. Limited information is available regarding cellular immune responses to vaccinia virus. We will obtain blood from vaccinated persons and measure immune responses in vi... | Upon review of all data

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Cohen, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Frey SE, Couch RB, Tacket CO, Treanor JJ, Wolff M, Newman FK, Atmar RL, Edelman R, Nolan CM, Belshe RB; National Institute of Allergy and Infectious Diseases Smallpox Vaccine Study Group. Clinical responses to undiluted and diluted smallpox vaccine. N Engl J Med. 2002 Apr 25;346(17):1265-74. doi: 10.1056/NEJMoa020534. Epub 2002 Mar 28. PMID 11923490
- [Background] Frey SE, Newman FK, Cruz J, Shelton WB, Tennant JM, Polach T, Rothman AL, Kennedy JS, Wolff M, Belshe RB, Ennis FA. Dose-related effects of smallpox vaccine. N Engl J Med. 2002 Apr 25;346(17):1275-80. doi: 10.1056/NEJMoa013431. Epub 2002 Mar 28. PMID 11923489
- [Background] Mathew A, Ennis FA, Rothman AL. Transient decreases in human T cell proliferative responses following vaccinia immunization. Clin Immunol. 2000 Aug;96(2):100-7. doi: 10.1006/clim.2000.4887. PMID 10900157
- [Derived] Cohen JI, Hohman P, Fulton R, Turk SP, Qin J, Thatcher K, Hornung RL. Kinetics of serum cytokines after primary or repeat vaccination with the smallpox vaccine. J Infect Dis. 2010 Apr 15;201(8):1183-91. doi: 10.1086/651453. PMID 20214479